CLINICAL TRIAL: NCT04445714
Title: A Prospective, Multicenter, Phase -IV Study to Assess the Safety of Fixed Dose Combination of Dapagliflozin and Saxagliptin in Indian Type 2 Diabetes Mellitus (T2D) Patients
Brief Title: To Assess Safety of Fixed Dose Combination of Dapagliflozin and Saxagliptin in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1683C00013
Record Dates: First submitted 2020-06-04; First posted 2020-06-24 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dapagliflozin and saxagliptin (Other): Singe arm once daily fixed dose combination of Dapa/Saxa 10 mg/5 mg administered orally
  Interventions: Drug: dapagliflozin and saxagliptin

INTERVENTIONS:
Drug: dapagliflozin and saxagliptin — Combination of dapagliflozin and saxagliptin tablet once daily fixed dose combination of Dapa/Saxa 10 mg/5 mg administered orally
  Other Names: QTERN Tablet

SUMMARY:
A prospective, multicenter, phase -IV study to assess the safety of fixed dose combination of dapagliflozin and saxagliptin in Indian Type 2 Diabetes Mellitus (T2D) patients.

DETAILED DESCRIPTION:
During the study, an AstraZeneca representative/delegate will have regular contacts with the study site, including visits to site for the site monitoring and source data verification activities. Electronic Case Report Forms (eCRF) will be used for data collection and query handling. The investigator will sign the completed electronic Case Report Forms. A copy of the completed electronic Case Report Forms will be archived at the study site. Authorized representatives of AstraZeneca or delegate, a regulatory authority, or an Ethics Committee may perform audits or inspections at the center's. Number and percentages of Incidence of adverse events will be presented, stratified by age/gender/baseline medications. Annualised event rate shall also be presented in addition to the incidence rate during the study. Mean change in HbA1C from baseline to 6 months for patients will be analysed using paired t test / Wilcoxon signed-rank test at 5% level of significance.

ELIGIBILITY:
Inclusion criteria:

For inclusion in the study subjects should fulfil the following criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures according to local Indian procedure.
2. Male and female patients aged > 18 and above
3. Documented history of type 2 diabetes mellitus with HbA1c level >7.0% and ≤ 10% at screening visit
4. Patients who are on a stable dose of antidiabetic drugs (including on Metformin dose between 1000-2000mg) in the past 3 months
5. Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent) to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.

Exclusion criteria:

1. Known allergies or contraindication to the contents of the IP, dapagliflozin or saxagliptin tablets.
2. Active participation in another clinical study with IP and/or investigational device
3. For women only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
4. Type 1 diabetes mellitus.
5. Treatment with a SGLT2 inhibitor, GLP-1 agonist or DPP4 inhibitors at Visit 1 or 2
6. Patients with moderate to severe renal impairment (eGFR persistently <45 mL/min/1.73 m2 by CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula or end-stage renal disease (ESRD) or 'Unstable or rapidly progressing renal disease
7. Patients with severe hepatic impairment (Child-Pugh class C)
8. History of pancreatitis or pancreatic surgery
9. Patients with a history of any malignancy
10. Patients with any of the following CV/Vascular Diseases within 3 months prior to signing the consent at enrolment, as assessed by the investigator:

    * Myocardial infarction.
    * Cardiac surgery or revascularization (CABG/PTCA).
    * Unstable angina.
    * Transient ischemic attack (TIA) or significant cerebrovascular disease.
    * Unstable or previously undiagnosed arrhythmia.
11. History of heart failure
12. Severe uncontrolled hypertension defined as systolic blood pressure ≥180 mm Hg and/or diastolic blood pressure ≥110 mm Hg at any visit up to randomisation
13. History of diabetic ketoacidosis
14. Any acute/chronic systemic infections
15. Recurrent urogenital infections
16. Patients at risk for volume depletion as judged by the investigator
17. Any condition which, in the judgment of the Investigator, may render the patient unable to complete the study or which may pose a significant risk to the patient or patient suspected or with confirmed poor protocol or medication compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Anil Bhansali, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Dr K P Singh, Principal Investigator — Fortis Hospital Mohali; Dr Indira Pattnaik, Principal Investigator — Sparsh Hospitals & Critical Care (P) Ltd, Bhubaneswar; Dr Sandeep Kumar Gupta, Principal Investigator — M V Hospital &Research centre Lucknow; Dr Faraz Farishta, Principal Investigator — Thumbay Hospital New Life Hyderabad; Dr Girithara Jayaram Naidu, Principal Investigator — KG Hospital
Locations (9):
- India (9):
  - Research Site, Bangalore
  - Research Site, Bhubaneswar
  - Research Site, Chandigarh
  - Research Site, Coimbatore
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Mohali
  - Research Site, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.'
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1683C00013&attachmentIdentifier=62fce152-e666-433a-82e6-a89b3b309b4f&fileName=Clinical_Study_Protocol_redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1683C00013&attachmentIdentifier=d5a753bc-2a19-48b3-aee3-130749ea1bed&fileName=Statistical_Analysis_Plan_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1683C00013&attachmentIdentifier=71ceea03-9bf6-4300-aeb0-70ffe7e45b5e&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg: All participants were given once daily fixed dose combination of Dapagliflozin 10 mg / Saxagliptin 5 mg administered orally at the same time of the day throughout the study.
Period: Overall Study
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Started | 196
Completed | 173
Not Completed | 23
Not completed — Discontinuation of the study | 14
Not completed — High plasma glucose-fasting and HbA1c; investigator decision to withdraw participant | 1
Not completed — Withdrawal of Informed Consent | 8

BASELINE CHARACTERISTICS:
Population: Enrolled population
Groups:
- Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mgOverall: All participants were given once daily fixed dose combination of Dapagliflozin 10 mg / Saxagliptin 5 mg administered orally at the same time of the day throughout the study.
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mgOverall
Number analyzed (Participants) | 196
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 196
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeters] | 163 (8.62)
Weight [Mean (Standard Deviation); unit: kilograms] | 74.2 (12.59)
Waist circumference [Mean (Standard Deviation); unit: centimeters] | 97.5 (12.76)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (4.35)
Glycated haemoglobin [Mean (Standard Deviation); unit: percentage of glycated haemoglobin] | 8.6 (0.77)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 161.8 (52.30)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data only available for 151 participants
  mmHg
    number analyzed (Participants) | 151
    (all) | 125.7 (9.27)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) Including Serious Adverse Events (SAEs), AEs Leading to Discontinuation (DAE), and Adverse Events of Special Interest
Description: Adverse events (AEs) including serious adverse events (SAEs), AEs leading to discontinuation (DAE), and adverse events of special interest (volume depletion, renal events, major hypoglycemic events, fractures, urinary/genital tract infections diabetic ketoacidosis, amputations and hospitalization for heart failure)
Time Frame: Baseline to End of Study (Week 26)
Population: Safety Population
Measure: Number; unit: events
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
events
  AEs | 40
  SAEs | 0
  DAEs | 0
  Adverse events of special interest | 4

2. Primary Outcome: Clinically Important or Significant Abnormalities in Safety Laboratory Values
Description: Clinical laboratory results were presented separately for haematology, clinical chemistry, and urinalysis variables.
  The number of participants with clinically important (haematology and clinical chemistry) or clinically significant (urinalysis) abnormalities in safety laboratory values are presented.
Time Frame: Enrolment (Week -1) to End of Study (Week 26)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
Participants | 0

3. Primary Outcome: Clinically Important Abnormalities in ECG Values
Description: The number of participants with clinically important abnormalities in ECG values are presented.
Time Frame: Time Frame: Baseline to End of Study (Week 26)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
Participants | 0

4. Primary Outcome: Clinically Important Abnormalities in Vital Signs (Pulse and Blood Pressure)
Description: The number of participants with clinically important abnormalities in vital signs (pulse and blood pressure).
Time Frame: Enrolment (Week -1) to End of Study (Week 26)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
Participants | 0

5. Primary Outcome: Clinically Significant Abnormalities in Physical Examinations
Description: The number of participants with clinically significant abnormalities in physical examinations.
Time Frame: Enrolment (Week -1) to End of Study (Week 26)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
Participants | 0

6. Secondary Outcome: Glycated Haemoglobin (HbA1c) Change at Week 24 Compared to Baseline
Description: The efficacy of the fixed dose combination of dapagliflozin + saxagliptin in Indian Type 2 Diabetes Mellitus participants was analyzed by measuring HbA1c change at week 24 compared to baseline.
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of glycated haemoglobin
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
percentage of glycated haemoglobin
  Baseline (Visit 2) | 8.6 (0.77)
  Week 24: number analyzed (Participants) | 189
  Week 24 | 7.4 (0.98)
  Change from Baseline: number analyzed (Participants) | 189
  Change from Baseline | -1.2 (1.09)
Statistical Analysis 1: Comparison: Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg; Change from baseline; Test type: Superiority; p < .0001, Paired t-test test; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.34 to -1.03]

7. Secondary Outcome: Weight Change at Week 24 Compared to Baseline
Description: The efficacy of the fixed dose combination of dapagliflozin + saxagliptin in Indian Type 2 Diabetes Mellitus participants was analyzed by measuring weight change at week 24 compared to baseline.
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
kilograms
  Baseline (Visit 2) | 74.2 (12.59)
  Week 24: number analyzed (Participants) | 189
  Week 24 | 72.2 (11.51)
  Change from Baseline: number analyzed (Participants) | 189
  Change from Baseline | -2.1 (3.98)
Statistical Analysis 1: Comparison: Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg; Change from baseline; Test type: Superiority; p < .0001, Paired t-test test; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-2.66 to -1.51]

8. Secondary Outcome: Systolic Blood Pressure Change at Week 24 Compared to Baseline
Description: The efficacy of the fixed dose combination of dapagliflozin + saxagliptin in Indian Type 2 Diabetes Mellitus participants was analyzed by measuring systolic blood pressure change at week 24 compared to baseline.
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
mmHg
  Baseline (Visit 2): number analyzed (Participants) | 151
  Baseline (Visit 2) | 125.7 (9.27)
  Week 24: number analyzed (Participants) | 189
  Week 24 | 124.5 (10.33)
  Change from Baseline: number analyzed (Participants) | 144
  Change from Baseline | -0.2 (12.90)
Statistical Analysis 1: Comparison: Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg; Change from baseline; Test type: Superiority; p = 0.8416, Paired t-test test; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.34 to 1.91]

9. Secondary Outcome: Fasting Plasma Glucose Change at Week 24 Compared to Baseline
Description: The efficacy of the fixed dose combination of dapagliflozin + saxagliptin in Indian Type 2 Diabetes Mellitus participants was analyzed by measuring fasting plasma glucose change at week 24 compared to baseline.
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
Number analyzed (Participants) | 196
mg/dL
  Baseline (Visit 2) | 161.8 (52.30)
  Week 24 | 136.7 (41.98)
  Change from Baseline | -24.4 (62.89)
Statistical Analysis 1: Comparison: Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg; Change from baseline; Test type: Superiority; p < .0001, Paired t-test test; Mean Difference (Final Values) = -24.4, 95% CI 2-sided [-33.4 to -15.4]

ADVERSE EVENTS:
Time Frame: Week 0 to End of Study (26 weeks)
Description: An adverse event was any unfavourable and unintended sign (e.g. an abnormal laboratory finding), symptom (for example nausea, chest pain), or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg
All-Cause Mortality (participants affected / at risk) | 0/196
Serious Adverse Events (participants affected / at risk) | 0/196
Other Adverse Events (participants affected / at risk) | 22/196
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed Dose Combination of Dapagliflozin 10 mg / Saxagliptin 5 mg (N=196)
Hypersensitivity (Immune system disorders) | 1 (1)
Balanitis candida (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Trichomoniasis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (7)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of or make presentations related to the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT04445714/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04445714/SAP_001.pdf